CLINICAL TRIAL: NCT03918980
Title: A 6-part First-in-human Study of LOU064 Consisting of a 4-part Randomized, Double-blind, Placebo-controlled SAD and MAD Study to Investigate the Safety and Tolerability in Healthy Volunteers, Subjects With Atopic Diathesis and Subjects With Atopic Dermatitis, an Open-label Food Effect Study and a Double-blind Formulation Effect Study in Healthy Volunteers
Brief Title: Single Dose and Multiple Dose Study to Assess Safety and Tolerability of LOU064
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOU064X2101
Record Dates: First submitted 2015-12-14; First posted 2019-04-18 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers, Atopic Diathesis and Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (27):
- Part 1 Dose A (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose B (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose C (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose D (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose E (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose F (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose G (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose H (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose I (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Dose J (Experimental): (Single Ascending Dose) Healthy volunteers will receive a single dose of LOU064.
  Interventions: Drug: LOU064
- Part 1 Placebo (Placebo Comparator): (Single Ascending Dose) Healthy volunteers will receive a single dose of placebo.
  Interventions: Drug: Placebo
- Part 2 Dose K (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Dose L (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Dose M (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Dose N (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Dose O (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Dose P (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 once daily for 12 days
  Interventions: Drug: LOU064
- Part 2 Placebo (Placebo Comparator): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take placebo once daily for 12 days
  Interventions: Drug: Placebo
- Part 3 Dose Fasted (Experimental): Healthy volunteers will receive a single dose of LOU064 given under fasting conditions followed by a single dose of LOU064 given after a high fat meal (cross-over design).
  Interventions: Drug: LOU064
- Part 3 Dose Fed (Experimental): Healthy volunteers will receive a single dose of LOU064 given after a high fat meal followed by a single dose of LOU064 given under fasting conditions (cross-over design).
  Interventions: Drug: LOU064
- Part 4 Dose R (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 twice daily for 12 days
  Interventions: Drug: LOU064
- Part 4 Dose S (Experimental): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take LOU064 twice daily for 12 days
  Interventions: Drug: LOU064
- Part 4 Placebo (Placebo Comparator): (Multiple Ascending Dose) Healthy Volunteers with asymptomatic atopic diathesis will take placebo twice daily for 12 days
  Interventions: Drug: Placebo
- Part 5 Formulation A (Experimental): Healthy Volunteers will receive a single dose of LOU064 formulation A followed by a single dose of LOU064 formulation B (cross-over design).
  Interventions: Drug: LOU064
- Part 5 Formulation B (Experimental): Healthy Volunteers will receive a single dose of LOU064 formulation B followed by a single dose of LOU064 formulation A (cross-over design).
  Interventions: Drug: LOU064
- Part 6 Dose T (Experimental): Subjects with atopic dermatitis will receive a twice daily dose of LOU064 for 4 weeks
  Interventions: Drug: LOU064
- Part 6 Placebo (Placebo Comparator): Subjects with atopic dermatitis will receive a twice daily dose of placebo for 4 weeks
  Interventions: Drug: LOU064; Drug: Placebo

INTERVENTIONS:
Drug: LOU064 — LOU064 will be administered as oral capsules in parts 1 to 6.
  Arms: Part 1 Dose A; Part 1 Dose B; Part 1 Dose C; Part 1 Dose D; Part 1 Dose E; Part 1 Dose F; Part 1 Dose G; Part 1 Dose H; Part 1 Dose I; Part 1 Dose J; Part 2 Dose K; Part 2 Dose L; Part 2 Dose M; Part 2 Dose N; Part 2 Dose O; Part 2 Dose P; Part 3 Dose Fasted; Part 3 Dose Fed; Part 4 Dose R; Part 4 Dose S; Part 5 Formulation A; Part 5 Formulation B; Part 6 Dose T; Part 6 Placebo
Drug: Placebo — Matching placebo capsules will be administered in parts 1,2, 4 and 6.
  Arms: Part 1 Placebo; Part 2 Placebo; Part 4 Placebo; Part 6 Placebo

SUMMARY:
This is a 6-part first-in-human study in up to approximately 184 participants. Parts 1 to 5 is in health volunteers and part 6 is in subjects with atopic dermatitis.

The purpose of this first-in-human study is to assess the safety and tolerability and pharmacokinetics (PK) of single and multiple doses of LOU064 both as once and twice daily oral administration in healthy volunteers and those with atopic diathesis or atopic dermatitis. This study will also explore the effect of food intake and different drug substance particle sizes on the in vivo disposition of LOU064 in healthy volunteers to guide dosing and formulation development for future clinical trials.

The study is registered on CT.Gov with the initiation of part 6 in patients (FPFV in April 2019).

DETAILED DESCRIPTION:
The study is composed of the following parts:

Part 1 is a double-blind, placebo-controlled single ascending dose (SAD) escalation study of up to 10 cohorts (N = approximately 80) in healthy volunteers Part 2 is a double-blind, placebo-controlled multiple ascending dose (MAD) escalation study in up to 6 cohorts in healthy volunteers with asymptomatic atopic diathesis with a 12-day treatment period (daily dosing) and 4-day follow-up period (N = approximately 48) Part 3 is a single cohort, single dose, open-label crossover food effect study (N = approximately 12) in healthy volunteers Part 4 is a double-blind, placebo-controlled multiple dose study in up to 2 cohorts of healthy volunteers with asymptomatic atopic diathesis with a 12-day treatment period (twice daily dosing) and 4-day follow-up period (N = approximately 16) Part 5 is a double-blind, single dose, crossover formulation effect study (N = approximately 12) in healthy volunteers Part 6 is a double-blind, placebo-controlled multiple dose study in subjects with atopic dermatitis with a 4-week treatment period (twice daily dosing of LOU064) and 3-week follow-up period in approximately 16 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female healthy subjects with an age range between 18 and 65 years (inclusive), and in good general health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening. Healthy subjects to participate in Part 2 or Part 4 must additionally have an atopic diathesis to be eligible for these specific study portions. Atopic healthy volunteers must have a positive skin prick test to a known allergen at screening (atopic diathesis) but must be clinically asymptomatic and not requiring any systemic medication. To participate in Part 6, subjects must additionally have chronic atopic dermatitis (AD) according to American Academy of Dermatology Consensus Criteria (Eichenfield et al 2014), that has been present for at least 1 year before the baseline visit and defined as:

   * Eczema Area and Severity Index (EASI) ≥ 12 at screening and baseline
   * IGA (Investigator's Global Assessment) ≥ 3 on a 5-point scale at screening and baseline
   * BSA (Body Surface Area) involvement ≥ 8% at screening and baseline
   * Subjects have applied a stable dose of bland topical emollient at least twice daily for at least 7 consecutive days immediately before the baseline visit
3. Able to communicate well with the Investigator, to understand and comply with the requirements of the study.
4. Subjects must weigh at least 50 kg and must have a body mass index (BMI) within the range of 18 -30 kg/m2 (inclusive) (parts 1-5) / 18-35 kg/m2 inclusive (part 6). BMI = body weight (kg) / [Height (m)]2.
5. At screening, and first baseline, vital signs (body temperature, systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three minutes and again (when required) after three minutes in the standing position. Sitting vital signs should be within the following ranges (inclusive):

   * Oral body temperature between 35.0-37.5 °C
   * Systolic blood pressure 90-139 mm Hg; for subjects ≥ 55 years, systolic blood pressure up to 149 mm Hg is accepted (part 6)
   * Diastolic blood pressure 50-89 mm Hg
   * Pulse rate 50 - 90

Exclusion Criteria

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Known family history or known presence of long QT syndrome.
4. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening and/or pre-treatment: PR > 200 msec QRS complex > 120 msec QTcF > 450 msec (males) QTcF > 460 msec (females)
5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
6. Known history of or current clinically significant arrhythmias.
7. Use of any systemic prescription drugs (including CYP3A inducers and inhibitors, and drugs with arrhythmogenic potential) other than hormonal contraceptives for women of childbearing potential, herbal supplements, within four (4) weeks prior to initial dosing or within 3 months for biologics (like dupilumab), and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing. If needed, (i.e. an incidental and limited need) paracetamol is acceptable, but must be documented in the Concomitant medications / Significant non-drug therapies page of the eCRF.

   For topical treatments in Part 6, the following rules apply:
   * Topical corticosteroids (TCS) and topical calcineurin inhibitors (TCI) must be stopped

     1 week prior to randomization to allow an adequate washout-period.
   * Other topical treatments for AD such as crisaborole, tar etc. and prescription moisturizers or moisturizers containing ingredients such as ceramides, lactic acid, urea, α-hydroxy- or fruit acids, vitamins A, D or E must be discontinued during the 4-week treatment period.
   * Phototherapy or tanning booth treatment must have stopped 4 weeks prior to baseline.
8. Donation or loss of 400 mL or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
10. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 7 days after stopping LOU064. Highly effective contraception methods include:

    - Total abstinence (when this is in line with the preferred and usual lifestyle of the subject.

    Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
    * Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
11. Hemoglobin levels below 12.0 g/dL at screening or first baseline.
12. Platelet count outside of the normal range (below 150x109/L or above 450 x 109) at screening or first baseline.
13. Significant illness that has not resolved within two (2) weeks prior to initial dosing.
14. Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
15. Recent (within the last three years (parts 1-5)/ within the last year (part 6)) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease requiring moderate to high dose systemic steroid medication (oral or parenteral).
16. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:

    * Inflammatory bowel disease, peptic ulcers, gastrointestinal including rectal bleeding.
    * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel Resection.
    * Pancreatic injury or pancreatitis.
    * Liver disease or liver injury as indicated by abnormal liver function tests. ALT (SGPT), AST (SGOT), γ-GT, alkaline phosphatase and serum bilirubin will be tested and need to be within the normal range at screening (parts 1-5) / must be within 1.5-fold of the upper limit of normal (ULN) at screening and assessed by the Investigator as not clinically significant (part 6).
    * If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to randomization, to rule out laboratory error.
    * History or presence of impaired renal function as indicated by clinically significantly
    * abnormal creatinine or BUN and/or urea values, or abnormal urinary constituents (e.g. albuminuria).
    * Evidence of urinary obstruction or difficulty in voiding at screening.
17. Flu-like symptoms within two weeks prior to dosing.
18. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
19. A positive Hepatitis B test result (Hepatitis B surface antigen/Hepatitis B core antibody) or Hepatitis C test result.
20. Subjects with a latent TB infection as indicated by the absence of any signs of active TB disease but with a positive IGRA.
21. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening and/or first baseline.
22. Any clinically significant white blood cell count or clinically significant white blood cell lab abnormalities at screening and/or baseline.
23. Any clinically significant abnormalities in any of the standard coagulation tests including the prothrombin time (PT), partial thromboplastin time (PTT), or International Normalized Ratio (INR) at screening and/or baseline.
24. Active smokers or use of tobacco products in the previous 3 months (parts 1-5). Heavy smokers who normally consume more than 10 cigarettes a day (part 6). Urine cotinine levels will be measured during screening and at each baseline for all subjects. Smokers will be defined as any subject who reports tobacco use and/or who has a positive urine cotinine level determined by local lab.
25. History or presence of any significant coagulation disorder, such as thrombocytopenia, hemophilia, or history of severe bleeding events, such as gastrointestinal (as evidenced by blood in stool) or subarachnoidal bleeding or recurrent spontaneous bleeding.
26. History or presence of thrombotic or thromboembolic event, or increased risk for thrombotic or thromboembolic event.
27. History or presence of cytopenia or bone marrow failure.
28. History or presence of poorly controlled asthma or asthma exacerbation as defined by worsening signs and symptoms prompting a medical intervention within the past 30 days.

    Subjects with asthma must have well-controlled disease as evidenced by use of rescue beta agonists no more than twice a week (except for relief of exercise-induced asthma) and wakening with nocturnal asthma no more than twice a month.
29. Any use of acetylsalicylic acid (ASA), COX-1 inhibitors, any other platelet inhibitors, or anticoagulants (e.g. warfarin) within two weeks prior to enrollment, including low dose ASA for prophylactic purposes.
30. History or presence of coronary artery disease, stroke, or transient ischemic attacks.
31. Polysorbate allergy or positive skin test for sensitivity to Tween 20 (i.e. score of "++" or greater).
32. History or presence of malignancy or obligatory precancerous condition of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
33. Sexually active males must use a condom during intercourse while taking drug and for 7 days after stopping study medication and should not father a child in this period.

    A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
34. Live vaccine (this includes nasal-spray flu vaccination) from 6 weeks prior to screening up to 7 days after the last study drug administration.
35. Vulnerable subjects, e.g. subjects kept in detention, soldiers, employees of the sponsor or a clinical research organization, involved in this study.
36. Subjects previously enrolled and dosed in any part of this study are not eligible to re-enroll in the same or another part

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part 1: 22 days, Part 2: 33 days, Part 3: 40 days, Part 4: 33 days, Part 5: 26 days, Part 6: 50 days
  Clinically significant changes in physical examination and anamnesis, vital signs, ECG, safety laboratory will be reported under (S)AEs.

SECONDARY OUTCOMES:
LOU064 pharmacokinetics Cmax | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  Cmax:The observed maximum plasma (or serum or blood) concentration following drug administration [mass / volume]
LOU064 pharmacokinetics Tmax | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  Tmax: The time to reach the maximum concentration after drug administration [time]
LOU064 pharmacokinetics AUCinf | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  AUCinf: The area under the plasma (or serum or blood) concentration-time curve from time zero to infinity [mass x time / volume]
LOU064 pharmacokinetics AUClast | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  AUClast: The area under the plasma (or serum or blood) concentration-time curve from time zero to the time of the last quantifiable concentration [mass x time / volume]
LOU064 pharmacokinetics AUCtau | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  AUCtau: The area under the plasma (or serum or blood) concentration-time curve from time zero to the end of the dosing interval tau [mass x time / volume]
LOU064 pharmacokinetics T1/2 | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  T1/2: The terminal elimination half-life [time]
LOU064 pharmacokinetics CL/F | Part 1: Day 1, 2, 3, 4, 5 and 8, Part 2: Day 1, 2, 3, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 3: Day 1, 2, 3, 4 and 5, Part 4: Day 1, 2, 3, 4, 5, 7, 9, 12, 13, 14, 15, 16 and 19, Part 5: Day 1, 2, 3, 5 and 8 Part 6: Day 1, 2, 8, 15, 22, 29, and day 30
  CL/F: The apparent systemic (or total body) clearance from plasma (or serum or blood) following extravascular administration [volume / time]

CONTACTS AND LOCATIONS:
Locations (2):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Leiden, Netherlands

REFERENCES:
- See also: Results for CLOU064X2101 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17793
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=719